CLINICAL TRIAL: NCT05362201
Title: Application of the Visualization of Treatment Objective (VTO) Analyses in the Treatment of the Temporomandibular Joint Disc Displacement
Brief Title: Application of the Visualization of Treatment Objective (VTO) Analyses in Fabricating Anterior Repositioning Splints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Hao Yu, Fujian Medical University, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20220309
Record Dates: First submitted 2022-04-15; First posted 2022-05-05 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Temporomandibular Joint Disorders
Keywords: temporomandibular Joint Anterior Disc Displacement; the visualization of treatment objective (VTO); anterior repositioning Splint
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: A randomised clinical trial was conducted with 20 patients diagnosed with ADDWR through RDC/TMD and they were randomly allocated into the group 1(traditional group):the therapeutic position of the ARS were determinded by the "minimum protrusive position";group2(digitial group): the therapeutic position of the ARS were determinded by the VTO analyse.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the therapeutic position of the ARS were determinded by the "minimum protrusive position" (Active Comparator): the therapeutic position of the ARS were determinded by the "minimum protrusive position",which was the traditional method to fabricate the anterior repositioning splints,the patients were instructed to protrusive the mandible in a therapeutic position in which the click is eliminated.
  Interventions: Procedure: therapeutic position of the anterior repositioning splints
- the therapeutic position of the ARS were determinded by the VTO analyse (Experimental): the therapeutic position of the ARS were determinded by the VTO analyse,first,the participants were constructed to take CBCT and MRI scans,the ideal therapeutic position of the ARS were located in which the temporomandibular joint space distribute well and the condylar recapture the disc,the dentist could determine the amount of condylar movement and performed VTO analyse by assessing the CBCT and MRI scans ,then it could easily realize the final condylar movements with the application of the dental articulator.
  Interventions: Procedure: therapeutic position of the anterior repositioning splints

INTERVENTIONS:
Procedure: therapeutic position of the anterior repositioning splints — the ADDWR paricipants will be allocated into 2 grounps and treated with anterior repositioning splints determined by traditional and digitial method respectively.

SUMMARY:
This study conducted a randomized controlled clinical trial to evaluate the effect of the the therapeutic position of the anterior repositioning splint determined by VTO analyse compared with traditional method for the treatment of the Anterior Disk Displacement with Reduction of the Temporomandibular Joint.

DETAILED DESCRIPTION:
A randomised clinical trial was conducted with 20 patients diagnosed with ADDWR through RDC/TMD and they were randomly allocated into the group 1(traditional group):the therapeutic position of the ARS were determinded by the "minimum protrusive position",which was the traditional method to fabricate the anterior repositioning splints;group2(digitial group): the therapeutic position of the ARS were determinded by the VTO analyse,first,the participants were constructed to take CBCT and MRI scans,the ideal therapeutic position of the ARS were located in which the temporomandibular joint space distribute well and the condylar recapture the disc,the dentist could determine the amount of condylar movement and performed VTO analyse by assessing the CBCT and MRI scans ,then it could easily realize the final condylar movements with the application of the dental articulator.

They were followed-up in the baseline,1 month,2 and 3 months after the inserted of the splints using the Craniomandibular Index (CMI) for temporomandibular joint function and PHQ-9,GAD-7 for psychological assessments,the tmj space and disc-condylar angle were measured through the CBCT and MRI scans,before and after ARS therapy.

ELIGIBILITY:
Inclusion Criteria:

* anterior disc displacement with reduction (ADDWR) confirmed by magnetic resonance imaging (MRI)
* Classified as ASA 1 or 2
* Willing to participate and sign a written informed consent form.

Exclusion Criteria:

* pregnant women
* heart pace disorders and epilepsy

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
temporomandibular joint function | up to three months
  the Craniomandibular Index (CMI) was used to assess the temporomandibular joint function after the inserted of the splints.

SECONDARY OUTCOMES:
psychological assessment the PHQ-9 | three months
  the PHQ-9 were used to assess the psychological factors in the baseline,1 month,2 and 3 months after the inserted of the splints.
psychological assessment GAD-7 | three months
  GAD-7 were used to assess the psychological factors in the baseline,1 month,2 and 3 months after the inserted of the splints.
disc-condyle angle | three months
  the disc-condyle angle were measured through MRI scan
temporomandibular joint space | three months
  the temporomandibular joint space were calculated through CBCT scan

CONTACTS AND LOCATIONS:
Overall Officials: Hao Yu, Principal Investigator — Fujian Medical University
Locations (1):
- Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No